CLINICAL TRIAL: NCT04308057
Title: Exploring the Effects of Aquatic Exercise on Cardiovascular Function in Older Adults
Acronym: ACELA
Status: Completed | Type: Observational
Sponsor: Sheffield Hallam University (Other)
Responsible Party: Sponsor
Other Study IDs: ER5320861
Record Dates: First submitted 2020-02-24; First posted 2020-03-13 (Actual); Last update posted 2022-09-15 (Actual); Status verified 2022-09

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Aquatic Therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Aquatic Exercise: General inclusion criteria included being over 55 years of age and normotensive (e.g., <140/90 mm Hg). Specifically for this group, we include participants engaging in swimming or other aquatic, primarily aerobic-based, training regimes for more than 2 times a week, for more than 6 months, at the time of the assessments.
- Land-based exercise: General inclusion criteria included being over 55 years of age and normotensive (e.g., <140/90 mm Hg). Specifically for this group, we include participants engaging in land-based, primarily aerobic training regimes (e.g. aerobic exercise) for more than 2 times a week, for a period longer than 6 months, at the time of the assessments.
- Mixed exercise: General inclusion criteria included being over 55 years of age and normotensive (e.g., <140/90 mm Hg). Specifically for this group, we include participants engaging in both land-based and aquatic, primarily aerobic, exercise regimes on an equal basis, for more than 6 months.
- Sedentary.: General inclusion criteria included being over 55 years of age and normotensive (e.g., <140/90 mm Hg). Specifically for this group, we include participants who are sedentary (e.g., defined as undertaking less than 60 min of structured/planned physical activity per week), for a period longer than 6 months.
  Interventions: Procedure: Aquatic exercise

INTERVENTIONS:
Procedure: Aquatic exercise — Participants belonging to Group D (sedentary group) will be randomised 1-to-1 between remaining sedentary (n=20) and following a self-managed, 8-week, aquatic-based exercise programme (n=20). The latter group will be offered an 8-week access to pool facilities. For Group D participants, all baseline assessments will be repeated at 8 weeks.
  Groups: Sedentary.

SUMMARY:
Cardiovascular ageing is implicated in the development of cardiovascular disease (CVD). Aquatic exercise is being considered as a co-adjuvant form of rehabilitation, but there is limited evidence for its cardiovascular risk-reduction properties for older people. Our study aims to address this by exploring the cardiovascular effects of long-term aquatic exercise in older adults in comparison to those who are either inactive or engaged in land-based/mixed training by measurement of micro- and macro-circulation.

ELIGIBILITY:
Inclusion Criteria:

* being over 55 years of age and normotensive (e.g., <140/90 mm Hg).

Exclusion Criteria:

* any overt chronic disease which would affect microvascular functioning,
* anaemia (irrespective of whether an iron supplementation course is followed or not)
* a recent (3 months' ago) major surgery
* None of the participants were undertaking high intensity interval training of any form.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group A (n=20) consists of participants engaging in swimming or other aquatic, primarily aerobic-based, training regimes for more than 2 times a week, for more than 6 months, at the time of the assessments. Similarly, Group B (n=20) consists of participants engaging in land-based, primarily aerobic training regimes (e.g. aerobic exercise) for more than 2 times a week, for a period longer than 6 months, at the time of the assessments. Group C (n=20) consists of participants who were cengaging in both land-based and aquatic, primarily aerobic, exercise regimes on an equal basis, for more than 6 months, while Group D (n=40) consists of people who were sedentary (e.g., defined as undertaking less than 60 min of structured/planned physical activity per week), for a period longer than 6 months.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-02-19 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Nitric oxide-mediated, macro (arterial)- circulatory function. | Baseline.
  We will use FMD as a measure of endothelium-dependent, nitric oxide (NO)-mediated, macro (arterial)- circulatory function. Baseline scanning to assess resting vessel diameter will be recorded over 3 minutes, following a 10-minute resting period. A rapid inflation-deflation pneumatic cuff placed immediately distal to the elbow joint will be used to as an FMD stimulus.
Nitric oxide-mediated, macro (arterial)- circulatory function. | 8 weeks.
  We will use FMD as a measure of endothelium-dependent, nitric oxide (NO)-mediated, macro (arterial)- circulatory function. Baseline scanning to assess resting vessel diameter will be recorded over 3 minutes, following a 10-minute resting period. A rapid inflation-deflation pneumatic cuff placed immediately distal to the elbow joint will be used to as an FMD stimulus.

SECONDARY OUTCOMES:
Microcirculatory function | Baseline.
  Skin blood flow will be measured as cutaneous red blood cell flux using a Laser Doppler Flowmeter (LDF). Local thermal hyperaemia will be induced using a heating disc surrounding the probe. The probe will be attached to the skin using a double-sided adhesion sticker. Participants will be rested in a supine position in a temperature-controlled room with a constant ambient temperature of 24° C for 35 minutes. Heart rate and diastolic and systolic blood pressure was recorded from the left arm at 5-minute intervals throughout the protocol (Dinamap Dash 2500, GE Healthcare, USA). Baseline skin blood flow data will be recorded for 5 minutes with the local heating disc temperature set at 30° C. Following this, rapid local heating will be initiated to obtain maximal vasodilation and the temperature will be increased by 1° C every 10 seconds until 42° C was reached. This will then be maintained for 30 minutes following, which the test will be completed.
Microcirculatory function | 8 weeks.
  Skin blood flow will be measured as cutaneous red blood cell flux using a Laser Doppler Flowmeter (LDF). Local thermal hyperaemia will be induced using a heating disc surrounding the probe. The probe will be attached to the skin using a double-sided adhesion sticker. Participants will be rested in a supine position in a temperature-controlled room with a constant ambient temperature of 24° C for 35 minutes. Heart rate and diastolic and systolic blood pressure was recorded from the left arm at 5-minute intervals throughout the protocol (Dinamap Dash 2500, GE Healthcare, USA). Baseline skin blood flow data will be recorded for 5 minutes with the local heating disc temperature set at 30° C. Following this, rapid local heating will be initiated to obtain maximal vasodilation and the temperature will be increased by 1° C every 10 seconds until 42° C was reached. This will then be maintained for 30 minutes following, which the test will be completed.
Anthropometry - 1 | Baseline.
  Stature, waist and hip circumferences will be measured (all in cms).
Anthropometry - 2 | Baseline.
  Body mass will be measured.
Anthropometry - 1 | 8 weeks.
  Stature, waist and hip circumferences will be measured (all in cms).
Anthropometry - 2 | 8 weeks.
  Body mass will be measured.
EQ-5D-5L | Baseline.
  The EQ5D-5L questionnaire will be completed, to support assessment of quality of life.
EQ-5D-5L | 8 weeks.
  The EQ5D-5L questionnaire will be completed, to support assessment of quality of life.
SF-IPAQ | Baseline.
  The SF-IPAQ questionnaire will be completed, to assess physical activity levels.
SF-IPAQ | 8 weeks.
  The SF-IPAQ questionnaire will be completed, to assess physical activity levels.
Q-Risk | Baseline.
  The online Q-Risk questionnaire will be competed, which assesses the risk of cardiovascular disease risk
Q-Risk | 8 weeks.
  The online Q-Risk questionnaire will be competed, which assesses the risk of cardiovascular disease risk
Feasibility outcome - 1 | Baseline
  Recruitment rate (% of those expressing an interest, being actually recruited).
Feasibility outcome - 2 | 8 weeks
  Adherence rate (% of those recruited completing at least 75% of the prescribed number of exercise sessions).
Feasibility outcome - 3 | 8 weeks
  Retention rate (% of those recruited completing the post-intervention assessments).

CONTACTS AND LOCATIONS:
Overall Officials: Markos Klonizakis, D.Phil., Principal Investigator — Sheffield Hallam University
Locations (1):
- Sheffield Hallam University, Sheffield, Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Ethical approval prevents data sharing.